CLINICAL TRIAL: NCT05023135
Title: DeepView SnapShot Portable (DV-SSP): Device Training Study
Status: Completed | Type: Observational
Sponsor: SpectralMD (Industry)
Responsible Party: Sponsor
Other Study IDs: CT-2021-01--CSP-10
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Burns; Wound Heal
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Subjects with Thermal Burn Injury: An initial imaging with the DV-SSP would be completed at the Study Site within 72 hours of suffering a thermal burn injury.
  Interventions: Device: DeepView SnapShot Portable (DV-SSP)

INTERVENTIONS:
Device: DeepView SnapShot Portable (DV-SSP) — DV-SSP assistive imaging to collect observational data

SUMMARY:
The purpose of this study is to continue development and validation of an algorithm for burn healing assessment by the Spectral MD DeepView device and provide burn healing potential assessment.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent or have a Legally Authorized Representative (LAR) able to do so;
* Life expectancy > 6 months;
* Thermal burn mechanism (flame, scald, or contact);
* The Study Burn(s) occurred less than 72 hours prior to the time of first imaging; and
* Minimum burn wound size for adult or pediatric patients is 0.5% TBSA per region
* For adult Subjects: Have 2 - 4 regions of their clinical burn(s) that meet the criteria for a Study Burn.
* For pediatric Subjects: Have 1 - 4 regions of their clinical burn(s) that meet the criteria for a Study Burn

Exclusion Criteria:

* Burn pattern distribution isolated to head, face, neck, hands, feet, genitalia, and/or joints;
* Subject has burns involving > 50% total body surface area (TBSA);
* Sepsis at the time of enrollment;
* Immunosuppression/radiation/chemotherapy < 3 months prior to enrollment;
* Concurrent use of investigational products with a known effect on the burn sites; and/or
* Any condition that in the opinion of the Investigator may prevent compliance with the study requirements or compromise subject safety.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects enrolled in this study will be recruited at the designated Study Site within 72 hours of suffering a thermal burn injury. Adult and pediatric Subjects with burns from one or more of the defined burn severities will be enrolled. All Subjects must meet the specified inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2023-04-09 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Predict area of severe burn, using measurement tools such as the Pearson Correlation Coefficient | 3 weeks
  Test that the Burn Segmentation Algorithm's predicted severe burn area (i.e., deep second degree and third degree) within an image of a burn injury, will be equivalent to the true area of severe burn as determined by the expert panel. The analysis for this study would only include data obtained from participants in the study.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Valleywise Health, Phoenix, Arizona
  - Bridgeport Hospital, Bridgeport, Connecticut
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Children's Hospital, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Stony Brook Medicine, Stony Brook, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - St. Christopher's Childrens Hospital, Philadelphia, Pennsylvania
  - University of South Carolina, Charleston, South Carolina